CLINICAL TRIAL: NCT04517721
Title: Effects of a Nurse-led Transitional Burns Rehabilitation Programme (4Cs-TBuRP) for Adult Burn Survivors at the Gansu Provincial Hospital, Lanzhou: A Randomised Controlled Trial
Brief Title: Effects of a Nurse-led Transitional Burns Rehabilitation Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Frances Kam Yuet WONG, Prof, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20200730001
Record Dates: First submitted 2020-08-14; First posted 2020-08-18 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Burns Multiple

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomised to either the control or intervention groups with the former receiving the existing care at the hospital and the latter receiving the both the new intervention and existing standard of care.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will receive same care at the pre-discharge phase. However in the post-discharge phase where participants are not likely to interact with each other, persons in the control group will continue to receive the usual care whilst persons in the treatment group receives the new intervention. The assigned group of participants will not be disclosed to the outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The 4C's-TBuRP for adult burn survivors comprises of two phases:
  * Phase 1: Discharge planning/ preparation and day of discharge (Comprehensive assessment and evaluation, Education, guidance, and counselling, Treatment and procedures, Case management (referral for nursing follow-up), multi-disciplinary follow-up and Surveillance)
  * Phase 2: Follow-up Phase (2 WeChat Telehealth, 6 structured telephone follow-ups and daytime patient/ family-initiated telephone service; home visit based on meeting criteria) over an 8-week follow-up with delivery of rehabilitation care across the spectrum by trained nurse case managers ongoing assessment, intervention using the Omaha System and delivery of evidence-based care.
  Interventions: Other: Nurse-Led Transitional Burns Rehabilitation Programme (4Cs-TBuRP)
- Control group (Active Comparator): Participants in the control group will receive the care at the discharge planning phase and thereafter continue to utilise the exiting service available at the hospital, that is, medical review in the hospital.
  Interventions: Other: Nurse-Led Transitional Burns Rehabilitation Programme (4Cs-TBuRP)

INTERVENTIONS:
Other: Nurse-Led Transitional Burns Rehabilitation Programme (4Cs-TBuRP) — The nurse-led transitional burns rehabilitation programme (4Cs-TBuRP) is presented as an 8-week interventional programme that supports holistic care for adult burn survivors led by a specialist burn care nurse and supported by the burn care team. The intervention posits that as the adult burn survivor transitions, several physiological, psychosocial, health-related behaviour and environmental needs emerge which lead to poor quality of life. Despite this, they may be unable to return to utilise available healthcare services or have inadequate contact with rehabilitation services. To facilitate their recovery and enhance the attainment of rehabilitation outcomes, the 4Cs-TBuRP views the burn care nurse as the link between rehabilitation services and the adult burn survivor. Thus, the burn care nurse serves as the coordinator of care and actively collaborates with the burn care team and the patient/ family to ensure that continuous care is delivered in a timely manner.

SUMMARY:
The number of adult burn survivors is increasing gradually, and attention is drawn towards how they can be supported during the transitioning period. Considering the impact of nurse-led programmes in chronic disease management, it is being argued that an appropriate nurse-led bridging transitional programme of care may be an essential extended/ add-on service for adult burn survivors. Guided by the Medical Research Council Framework for Complex Interventions, a nurse-led programme has been developed. This phase seeks to implement the intervention, evaluate its effects, and understand the mechanisms of implementation at the Gansu Provincial Hospital, Lanzhou.

A randomized controlled trial approach with a nested process evaluation phase will be used. Participants will be recruited from the Burn Unit of the Gansu Provincial Hospital, Lanzhou and the intervention commenced from at least 72 hours to discharge up to 2 months post-discharge. Participants will be randomized to either control or treatment group using a blinded approach. Following the completion of the intervention, up to 15 participants will be recruited for face to face interviews.

DETAILED DESCRIPTION:
Recovery following burn injury is a complex process which involves re-fitting one's new form into an already known world. The aftermath of burns and complex responses by affected persons makes it difficult to map a clear recovery pathway. At the initial phase of recovery, the patient may show several responses such as disbelief, fear, and pain. These responses may become more pronounced as the patient comes to terms with the losses associated with injury. Further challenges associated with appearance changes and function may accrue as healing progresses and the scars evolve through maturation. Subsequently by discharge, burn survivors need to adapt to a new situation as they return to the community and assume full responsibility of their care. Hospital discharge, therefore, does not imply an end to treatment but a transitional period when the burn patient is still coming to terms with the reality of the injury, identifying new approaches to thriving and adapting to the changes thereof. To facilitate this ongoing recovery of adult burn survivors, there is therefore a need for continuous contact with rehabilitation services to ensure that needs that emerge in the process are identified and actively resolved.

Considering the importance of rehabilitation in the recovery process of the adult burn patient, it becomes essential to ensure that all burn patients receive rehabilitative care as and when needed. However, burn rehabilitation practices vary across settings. In developed countries, the burn patients often undergo intensive rehabilitation concurrently with acute care and later stepped down to continue an inpatient rehabilitation programme before discharge. In contrast, burn centres in developing countries may not have such step down services to a unique inpatient rehabilitation service; thus, the patient benefits only from the rehabilitation service that occurs alongside acute care and thereafter discharged home. Pressure on beds and limited financial resources in some developing settings may also trigger early discharge from the burn unit which further shortens the patient's contact with rehabilitation services.

In Mainland China, the concept of rehabilitation is still under development, not commonly practiced and where available, burn patients may face limited access due to inadequate personnel. The escalating chronic disease burden and ageing population further leaves limited resources allocated to burns rehabilitation in Mainland China. Even in healthcare facilities with rehabilitation services, the cultural belief among Chinese citizens that rehabilitation is a natural outcome of diseases, rather than an active management of dysfunctional issues of the body may affect the level of service utilization. Previous studies in Mainland China have also highlighted the significant focus on medical management of burn injuries with limited attention to comprehensive rehabilitative support. Thus, at the time of discharge the adult burn survivors may not have received adequate rehabilitative support commensurate with their needs and have to live with serious disabilities.

As the adult burn survivor transitions from the hospital to the community, anxiety and uncertainties may ensue. Other emotional responses may become more pronounced as the adult burn survivor comes to terms with the injury and the losses associated with it. Thus, the adult burn survivor transitions to the early post-discharge period with several physical, psychological, and social needs whilst at the same time, they are expected to assume full responsibility for their care. By 3 months post-discharge, burn survivors experience increasing psychological burden, poor physical role performances and poor quality of life. Within 6 months to 1 year post-discharge without professional support, the adult burn patient may experience further emotional distress reflected by the high rates of depression, sleep disturbance, body image concerns and sexual problems. Although statistically insignificant, several studies have reported an improvement in burn-specific health beyond 1year post-burn. Besides, psychosocial distress may still persist by 9 years post-discharge. These strengthen the need for ongoing comprehensive and continuous care to facilitate early identification and resolution of biopsychosocial needs that may emerge; a care pathway similar to persons living with chronic conditions.

Along the recovery trajectory for adult burn survivors, findings from several studies suggest that the greatest physical and psychosocial decline may be experienced by 2-3 months post-discharge. This assertion implies that the discharge to early post-discharge period, that is, 2 months following discharge represent a vulnerable period which can impact adversely on the long-term recovery outcomes of adult burn survivors. The period has been described as unpredictable with the emergence of varied needs requiring an individualized approach to care on regular basis than is provided by interval outpatient clinic visits. Despite these assertions, it is around this period that professional support may be limited or unavailable and some adult burn survivors may not return to the hospital due to issues such as long travel distances and associated costs. These raise an interest regarding how professional support can be organized and delivered as the patient transitions to the early post-discharge period in the home or community to ensure that they receive the sustained and comprehensive rehabilitative support. Thus, the current study to develop a nurse-led transitional rehabilitation programme and evaluate its effects among adult burn survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years
2. Burn size ≥10% TBSA
3. Reachable on phone and WeChat
4. Absence of confirmed psychiatric condition
5. Absence of confirmed chronic diagnosis of renal failure or diabetes mellitus with foot ulcers

Exclusion Criteria:

Unable to communicate Not reachable via phone Confirmed underlying psychiatry or renal failure or diabetes mellitus with foot ulcers Already engaged in another burn rehabilitation programme Will not reside in the specified location within three months of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Simplified Chinese versions of Burn Specific Health Scale-Brief and the 5-level EQ-5D. | Three months
  The Burn Specific Health Scale-Brief comprises of 40 questions, 9 sub-scales, and 3 domains (physical, mental, and social). Each item is scored on a 5-point scale ranging from 0 (extremely) to 4 (not at all). The maximum score is 140. Lower scores suggest poor quality of life and higher scores imply good quality of life. Internal consistency of the total instrument has been reported to be α=0.94 with test-retest reliability suggesting that the Intraclass Correlation Coefficient (ICC) ranged from 0.81 to 0.96 with a total score of 0.93. The 5-level EQ-5D has five response levels: level 1 (no problem) to level 5 (extreme problem). The possible health states are defined by combining one level from each dimension. An EQ-5D-5L index value is calculated ranging from 0 (death) to 1 (full health). Decreasing scores therefore suggest poor health whilst increasing scores suggest good health.

SECONDARY OUTCOMES:
Chinese version of the Hospital Anxiety and Depression Scale | Three months
  The 14-item Hospital Anxiety and Depression Scale was designed as a tool to screen for anxiety and depressive symptoms in medical settings, and has well-demonstrated solid psychometric properties for use in medical settings and commonly used in burn care settings to screen anxiety and depression. The total score is 42 (21 per subscale). Scores per subscale can range from 0-21. Higher scores indicate greater levels of anxiety and depression and lower scores imply low levels of anxiety and depression.
Chinese version of the Pittsburgh Sleep Quality Index | Three months
  The Chinese version of the Pittsburgh Sleep Quality Index is a widely recognized instrument used to evaluate the quality of sleep. It includes 19 items with a total score that ranges from 0 to 21. A higher PSQI score implies poorer quality of sleep and lower scores imply good sleep patterns. In general, a PSQI score greater than 5 is considered to indicate poor sleep quality.
Chinese version of the Brief Pain Inventory | Three months
  : The Chinese version of the Brief Pain Inventory will be used to evaluate pain among participants. It has 15 items, of which 11 items have numeric rating scale, on the experience of pain, the area of severe pain, the presence of pain, minimum and maximum pain on the previous day, current pain level, analgesia and pain relief, and the interference of pain on the patient's functioning. Pain severity and interference scores are calculated out of a total score of 10. Higher scores represent increasing pain severity and interference.
Chinese version of a visual analogue scale | Three months
  The Chinese version of a visual analogue scale will be used to evaluate this itch intensity among participants. Intraclass correlation coefficient has been recorded as 0.88 (Reich et al., 2012). The tool ranges from 0 (no itch) to 10 (worst imaginable itch). Thus, increasing scores represent worsening itch.
Chinese version of the Disability of the Arm, Shoulder and Hand Symptom Scale (DASH) | Three months
  The DASH tool is a 30-item questionnaire that asks the patient to grade symptoms and physical function during the preceding week on a five-point Likert scale. The reliability of the DASH is excellent (intraclass correlation coefficient 0.97 with Cronbach's alpha of 0.97. The tool is scored from 0 (no disability) to 100. Increasing scores suggest the existence of a disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Gansu Provincial Hospital, Gansu, Lanzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albarran, J. (2005). Response to editorial: Nurse led care. British Medical Journal (BMJ), 330, 682-683.
- [Background] Brusselaers N, Monstrey S, Vogelaers D, Hoste E, Blot S. Severe burn injury in Europe: a systematic review of the incidence, etiology, morbidity, and mortality. Crit Care. 2010;14(5):R188. doi: 10.1186/cc9300. Epub 2010 Oct 19. PMID 20958968
- [Background] Chinese Burn Association; Chinese Association of Burn Surgeons; Cen Y, Chai J, Chen H, Chen J, Guo G, Han C, Hu D, Huan J, Huang X, Jia C, Li-Tsang CW, Li J, Li Z, Liu Q, Liu Y, Luo G, Lv G, Niu X, Peng D, Peng Y, Qi H, Qi S, Sheng Z, Tang D, Wang Y, Wu J, Xia Z, Xie W, Yang H, Yi X, Yu L, Zhang G; Chinese Burn Care and Rehabilitation Association. Guidelines for burn rehabilitation in China. Burns Trauma. 2015 Oct 21;3:20. doi: 10.1186/s41038-015-0019-3. eCollection 2015. PMID 27574666
- [Background] Christiaens W, Van de Walle E, Devresse S, Van Halewyck D, Benahmed N, Paulus D, Van den Heede K. The view of severely burned patients and healthcare professionals on the blind spots in the aftercare process: a qualitative study. BMC Health Serv Res. 2015 Aug 1;15:302. doi: 10.1186/s12913-015-0973-2. PMID 26231290
- [Background] Evers LH, Bhavsar D, Mailander P. The biology of burn injury. Exp Dermatol. 2010 Sep;19(9):777-83. doi: 10.1111/j.1600-0625.2010.01105.x. Epub 2010 Jul 14. PMID 20629737
- [Background] Gerber LH, Bush H, Holavanahalli R, Esselman P, Schneider J, Heinemann A, Garfinkel S, Cai C. A scoping review of burn rehabilitation publications incorporating functional outcomes. Burns. 2019 Aug;45(5):1005-1013. doi: 10.1016/j.burns.2018.09.029. Epub 2018 Oct 26. PMID 31203869
- [Background] Gullick JG, Taggart SB, Johnston RA, Ko N. The trauma bubble: patient and family experience of serious burn injury. J Burn Care Res. 2014 Nov-Dec;35(6):e413-27. doi: 10.1097/BCR.0000000000000030. PMID 25144806
- [Background] Hundeshagen G, Suman OE, Branski LK. Rehabilitation in the Acute Versus Outpatient Setting. Clin Plast Surg. 2017 Oct;44(4):729-735. doi: 10.1016/j.cps.2017.05.004. Epub 2017 Jul 28. PMID 28888298
- [Background] Jagnoor J, Lukaszyk C, Fraser S, Chamania S, Harvey LA, Potokar T, Ivers RQ. Rehabilitation practices for burn survivors in low and middle income countries: A literature review. Burns. 2018 Aug;44(5):1052-1064. doi: 10.1016/j.burns.2017.10.007. Epub 2017 Dec 28. PMID 29290511
- [Background] Kornhaber R, Rickard G, McLean L, Wiechula R, Lopez V, Cleary M. Burn care and rehabilitation in Australia: health professionals' perspectives. Disabil Rehabil. 2019 Mar;41(6):714-719. doi: 10.1080/09638288.2017.1406009. Epub 2017 Dec 5. PMID 29207887
- [Background] Lotfi M, Ghahremaneian A, Aghazadeh A, Jamshidi F. The Effect of Pre-Discharge Training on the Quality of Life of Burn Patients. J Caring Sci. 2018 Jun 1;7(2):107-112. doi: 10.15171/jcs.2018.017. eCollection 2018 Jun. PMID 29977882
- [Background] McAleavey AA, Wyka K, Peskin M, Difede J. Physical, functional, and psychosocial recovery from burn injury are related and their relationship changes over time: A Burn Model System study. Burns. 2018 Jun;44(4):793-799. doi: 10.1016/j.burns.2017.12.011. Epub 2018 Feb 1. PMID 29395409
- [Background] Procter F. Rehabilitation of the burn patient. Indian J Plast Surg. 2010 Sep;43(Suppl):S101-13. doi: 10.4103/0970-0358.70730. PMID 21321643
- [Background] Richmond TS, Thompson HJ, Deatrick JA, Kauder DR. Journey towards recovery following physical trauma. J Adv Nurs. 2000 Dec;32(6):1341-7. doi: 10.1046/j.1365-2648.2000.01629.x. PMID 11136401
- [Background] Schneider JC, Qu HD, Lowry J, Walker J, Vitale E, Zona M. Efficacy of inpatient burn rehabilitation: a prospective pilot study examining range of motion, hand function and balance. Burns. 2012 Mar;38(2):164-71. doi: 10.1016/j.burns.2011.11.002. Epub 2011 Nov 25. PMID 22119446
- [Background] Schneider JC, Mathews K, Ryan CM. Burn rehabilitation outcomes: lessons learned from the uniform data system for medical rehabilitation. J Burn Care Res. 2014 May-Jun;35(3):212-3. doi: 10.1097/BCR.0b013e318299d505. No abstract available. PMID 23799485
- [Background] Serghiou MA, Niszczak J, Parry I, Li-Tsang CWP, Van den Kerckhove E, Smailes S, Edgar D. One world one burn rehabilitation standard. Burns. 2016 Aug;42(5):1047-1058. doi: 10.1016/j.burns.2016.04.002. Epub 2016 May 5. PMID 27161089
- [Background] Sibbald RG, Ayello EA. Deep Burns: Comparing the Developed and Developing World. Adv Skin Wound Care. 2019 Jan;32(1):5. doi: 10.1097/01.ASW.0000550458.48419.d5. No abstract available. PMID 30570552
- [Background] Stylianou N, Buchan I, Dunn KW. A review of the international Burn Injury Database (iBID) for England and Wales: descriptive analysis of burn injuries 2003-2011. BMJ Open. 2015 Feb 27;5(2):e006184. doi: 10.1136/bmjopen-2014-006184. PMID 25724981
- [Background] Young AW, Dewey WS, King BT. Rehabilitation of Burn Injuries: An Update. Phys Med Rehabil Clin N Am. 2019 Feb;30(1):111-132. doi: 10.1016/j.pmr.2018.08.004. Epub 2018 Oct 31. PMID 30470416
- [Background] Askay SW, Stricklin M, Carrougher GJ, Patterson DR, Klein MB, Esselman PC, Engrav LH. Using QMethodology to identify reasons for distress in burn survivors postdischarge. J Burn Care Res. 2009 Jan-Feb;30(1):83-91. doi: 10.1097/BCR.0b013e3181921f42. PMID 19060733
- [Background] Barrett LW, Fear VS, Waithman JC, Wood FM, Fear MW. Understanding acute burn injury as a chronic disease. Burns Trauma. 2019 Sep 16;7:23. doi: 10.1186/s41038-019-0163-2. eCollection 2019. PMID 31534977
- [Background] Boeve SA, Aaron LA, Martin-Herz SP, Peterson A, Cain V, Heimbach DM, Patterson DR. Sleep disturbance after burn injury. J Burn Care Rehabil. 2002 Jan-Feb;23(1):32-8. doi: 10.1097/00004630-200201000-00007. PMID 11803310
- [Background] Cameron IM, Crawford JR, Lawton K, Reid IC. Psychometric comparison of PHQ-9 and HADS for measuring depression severity in primary care. Br J Gen Pract. 2008 Jan;58(546):32-6. doi: 10.3399/bjgp08X263794. PMID 18186994
- [Background] Chen J, Li-Tsang CW, Yan H, Liang G, Tan J, Yang S, Wu J. A survey on the current status of burn rehabilitation services in China. Burns. 2013 Mar;39(2):269-78. doi: 10.1016/j.burns.2012.06.016. Epub 2012 Sep 13. PMID 22981799
- [Background] Dowda DJ, Li F. Major concerns and issues in burn survivors in Australia. Burns Trauma. 2014 Apr 6;2(2):84-7. doi: 10.4103/2321-3868.130192. eCollection 2014. PMID 27602366
- [Background] Echevarría-Guanilo, M. E., Gonçalves, N., Farina, J. A., & Rossi, L. A. (2016). Assessment of health-related quality of life in the first year after burn. Escola Anna Nery, 20(1), 155-166.
- [Background] Ehde DM, Patterson DR, Wiechman SA, Wilson LG. Post-traumatic stress symptoms and distress following acute burn injury. Burns. 1999 Nov;25(7):587-92. doi: 10.1016/s0305-4179(99)00050-9. PMID 10563683
- [Background] Esselman PC, Askay SW, Carrougher GJ, Lezotte DC, Holavanahalli RK, Magyar-Russell G, Fauerbach JA, Engrav LH. Barriers to return to work after burn injuries. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S50-6. doi: 10.1016/j.apmr.2007.09.009. PMID 18036982
- [Background] Fauerbach JA, Lawrence JW, Munster AM, Palombo DA, Richter D. Prolonged adjustment difficulties among those with acute posttrauma distress following burn injury. J Behav Med. 1999 Aug;22(4):359-78. doi: 10.1023/a:1018726103302. PMID 10495968
- [Background] Knighton, J. (2020). Nursing Management of the Burn Patient. In Handbook of Burns Volume 1 (pp. 347-384): Springer.
- [Background] Lawrence JW, Fauerbach J, Eudell E, Ware L, Munster A. The 1998 Clinical Research Award. Sleep disturbance after burn injury: a frequent yet understudied complication. J Burn Care Rehabil. 1998 Nov-Dec;19(6):480-6. doi: 10.1097/00004630-199811000-00005. PMID 9848037
- [Background] Oster C, Willebrand M, Ekselius L. Burn-specific health 2 years to 7 years after burn injury. J Trauma Acute Care Surg. 2013 Apr;74(4):1119-24; discussion 1124. doi: 10.1097/TA.0b013e318283cca0. PMID 23511154
- [Background] Patterson DR, Everett JJ, Bombardier CH, Questad KA, Lee VK, Marvin JA. Psychological effects of severe burn injuries. Psychol Bull. 1993 Mar;113(2):362-78. doi: 10.1037/0033-2909.113.2.362. PMID 8451340
- [Background] Patterson DR, Ptacek JT, Cromes F, Fauerbach JA, Engrav L. The 2000 Clinical Research Award. Describing and predicting distress and satisfaction with life for burn survivors. J Burn Care Rehabil. 2000 Nov-Dec;21(6):490-8. PMID 11194801
- [Background] Roberts SB, Bonnici DM, Mackinnon AJ, Worcester MC. Psychometric evaluation of the Hospital Anxiety and Depression Scale (HADS) among female cardiac patients. Br J Health Psychol. 2001 Nov;6(Part 4):373-383. doi: 10.1348/135910701169278. PMID 12614511
- [Background] Serio-Melvin M, Yoder LH, Gaylord KM. Caring for burn patients at the United States Institute of Surgical Research: the nurses' multifaceted roles. Nurs Clin North Am. 2010 Jun;45(2):233-48. doi: 10.1016/j.cnur.2010.02.001. PMID 20510707
- [Background] Sveen J, Sjoberg F, Oster C. Health-related quality of life in Swedish pediatric burn patients and associations with burn and family characteristics. Burns. 2014 Aug;40(5):987-94. doi: 10.1016/j.burns.2013.10.005. Epub 2013 Nov 27. PMID 24290162
- [Background] Tang, D., Li-Tsang, C. W., Au, R. K., Li, K.-c., Yi, X.-f., Liao, L.-r., . . . Liu, C.-s. (2015). Functional outcomes of burn patients with or without rehabilitation in mainland China. Hong Kong journal of occupational therapy, 26(1), 15-23.
- [Background] Tang D, Li-Tsang CW, Au RK, Shen X, Li KC, Yi XF, Liao LR, Cao HY, Feng YN, Liu CS. Predictors of functional independence, quality of life, and return to work in patients with burn injuries in mainland China. Burns Trauma. 2016 Nov 4;4:32. doi: 10.1186/s41038-016-0058-4. eCollection 2016. PMID 27826591
- [Background] Van Loey NE, Van Son MJ. Psychopathology and psychological problems in patients with burn scars: epidemiology and management. Am J Clin Dermatol. 2003;4(4):245-72. doi: 10.2165/00128071-200304040-00004. PMID 12680803
- [Background] Wasiak J, Paul E, Lee SJ, Mahar P, Pfitzer B, Spinks A, Cleland H, Gabbe B. Patterns of recovery over 12 months following a burn injury in Australia. Injury. 2014 Sep;45(9):1459-64. doi: 10.1016/j.injury.2014.02.018. Epub 2014 Feb 20. PMID 24698152
- [Background] Wiechman SA, Ptacek JT, Patterson DR, Gibran NS, Engrav LE, Heimbach DM. Rates, trends, and severity of depression after burn injuries. J Burn Care Rehabil. 2001 Nov-Dec;22(6):417-24. doi: 10.1097/00004630-200111000-00012. PMID 11761394
- [Background] Wiechman SA, Carrougher GJ, Esselman PC, Klein MB, Martinez EM, Engrav LH, Gibran NS. An expanded delivery model for outpatient burn rehabilitation. J Burn Care Res. 2015 Jan-Feb;36(1):14-22. doi: 10.1097/BCR.0000000000000153. PMID 25198101
- [Background] Wiechman SA, McMullen K, Carrougher GJ, Fauerbach JA, Ryan CM, Herndon DN, Holavanahalli R, Gibran NS, Roaten K. Reasons for Distress Among Burn Survivors at 6, 12, and 24 Months Postdischarge: A Burn Injury Model System Investigation. Arch Phys Med Rehabil. 2018 Jul;99(7):1311-1317. doi: 10.1016/j.apmr.2017.11.007. Epub 2017 Dec 16. PMID 29258837
- [Background] Xia, Z.-Y., Kong, Y., Yin, T.-T., Shi, S.-H., Huang, R., & Cheng, Y.-H. (2014). The impact of acceptance of disability and psychological resilience on post-traumatic stress disorders in burn patients. International Journal of Nursing Sciences, 1(4), 371-375.
- [Background] Xiao Y, Zhao K, Ma ZX, Li X, Qiu YP. Integrated medical rehabilitation delivery in China. Chronic Dis Transl Med. 2017 Apr 29;3(2):75-81. doi: 10.1016/j.cdtm.2017.02.003. eCollection 2017 Jun 25. PMID 29063059
- [Derived] Bayuo J, Wong FKY, Wong AKC, Baffour PK, Chung LYF. A comprehensive nurse-led aftercare programme addressing post-burn sexual well-being of adult burn survivors: a randomised controlled trial. BMC Nurs. 2024 Nov 11;23(1):818. doi: 10.1186/s12912-024-02461-3. PMID 39529032
- [Derived] Bayuo J, Wong FKY, Chung LYF. Effect of a transitional tele-rehabilitation programme on quality of life of adult burn survivors: A randomised controlled trial. Clin Rehabil. 2024 Oct;38(10):1333-1345. doi: 10.1177/02692155241265930. Epub 2024 Aug 27. PMID 39191373
- [Derived] Bayuo J, Wong FKY, Chung LYF. Effects of a nurse-led transitional burns rehabilitation programme (4Cs-TBuRP) for adult burn survivors: protocol for a randomised controlled trial. Trials. 2021 Oct 13;22(1):698. doi: 10.1186/s13063-021-05679-7. PMID 34645512